CLINICAL TRIAL: NCT04803097
Title: Capsular Outcomes of Pediatric Cataract Surgery With Primary Intraocular Lens
Brief Title: Capsular Outcomes of Pediatric Cataract Surgery With Primary Intraocular Lens Implantation
Acronym: capsular
Status: Completed | Type: Observational
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: cataract- fuyana
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Capsular Contracture, Implant; Pediatric Cataract
Keywords: capsular outcome; pediatric cataract; posterior capsulorhexis
MeSH Terms: conditions — Implant Capsular Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric cataract group: Children who underwent cataract surgery and primary IOL implantation at the Eye Hospital of Wenzhou Medical University (Hangzhou, China) between 2016 and 2019 were included in the study. Every surgery included posterior capsulorhexis or capsulotomy and anterior vitrectomy. Patients accept slit-lamp-adapted anterior segmental photography at 1 week, 2 weeks, 1 month, 3 months, and 6 months postoperatively.

INTERVENTIONS:
Diagnostic Test:  — We took slit-lamp-adapted anterior segmental photography from pediatric cataract eyes at baseline，1 week, 2 weeks, 1 month, 3 months, and 6 months postoperatively.

SUMMARY:
Lens capsular often changes after pediatric cataract surgery，causing complications such as anterior capsulerhexis shrinkage, visual axis opacification (VAO), zonular dehiscence and so on. The aim of study was to prospectively investigate the capsular outcomes of pediatric cataract surgery with primary intraocular lens (IOL) implantation.

DETAILED DESCRIPTION:
To investigate the capsular outcomes from a case series of children who underwent cataract surgery and primary IOL implantation at the Eye Hospital of Wenzhou Medical University between 2016 and 2019. Took Digital retro-illumination photographs of pediatric eyes at baseline and 6 months, 12 months, and the last visit postoperatively. Compare the capsular outcomes of the posterior capsule opening (PCO) area and visual axis transparent area at those time points, and analysis the correlations between the PCO area and influential factors, such as age at surgery, axial growth, and follow-up duration.

ELIGIBILITY:
Inclusion Criteria:

Children (age 0.5~8 years) who underwent cataract surgery, posterior capsulorhexis or capsulotomy and anterior vitrectomyand primary IOL implantation at the Eye Hospital of Wenzhou Medical University (Hangzhou, China). The follow-up period was at least 1 year.

Exclusion Criteria:

Patients with ocular trauma, corneal disorders, glaucoma, preoperative lens luxation or subluxation, membranous cataract, persistent hyperplastic primary vitreous, surgical or postoperative complications such as glaucoma or suspect-glaucoma and synechia, pupils that could not be sufficiently dilated, and those who could not complete follow-ups or did not have clear digital photographs.

Ages: 6 Months to 96 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients （age：0.5~8.0 years）with congenital cataract
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
PCOA | 20.74 ± 7.89 months
  A comparison of posterior capsular opening areas at the corresponding time points
VATA | 20.74 ± 7.89 months
  A comparison of visual axis transparent areas at the corresponding time points

SECONDARY OUTCOMES:
axial length growth | 20.74 ± 7.89 months
  The growth of axial length at the corresponding time points

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] Lin H, Tan X, Lin Z, Chen J, Luo L, Wu X, Long E, Chen W, Liu Y. Capsular Outcomes Differ with Capsulorhexis Sizes after Pediatric Cataract Surgery: A Randomized Controlled Trial. Sci Rep. 2015 Nov 5;5:16227. doi: 10.1038/srep16227. PMID 26537991
- [Background] Tan X, Lin H, Lin Z, Chen J, Tang X, Luo L, Chen W, Liu Y. Capsular Outcomes After Pediatric Cataract Surgery Without Intraocular Lens Implantation: Qualitative Classification and Quantitative Measurement. Medicine (Baltimore). 2016 Mar;95(10):e2993. doi: 10.1097/MD.0000000000002993. PMID 26962807
- [Derived] Fu Y, Wang D, Ding X, Chang P, Zhao Y, Hu M, Li Z, Zhao YE. Posterior Capsular Outcomes of Pediatric Cataract Surgery With In-The-Bag Intraocular Lens Implantation. Front Pediatr. 2022 Apr 8;10:827084. doi: 10.3389/fped.2022.827084. eCollection 2022. PMID 35463896